CLINICAL TRIAL: NCT06202742
Title: Effects of Cognitive Behavioral Therapy for Insomnia in Type 2 Diabetes Mellitus: A Randomized Controlled Trial
Brief Title: Cognitive Behavioral Therapy for Insomnia in Type 2 Diabetes Mellitus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MURA2023/873
Record Dates: First submitted 2023-12-12; First posted 2024-01-11 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Type 2 Diabetes; Insomnia
Keywords: cognitive behavioral therapy for insomnia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive behavioral therapy (Experimental): Cognitive behavioral therapy for insomnia (CBTI) is non-medical treatment to improve insomnia. CBTI group will attend online meeting, 1 hour weekly for 8 weeks.
  Interventions: Behavioral: cognitive behavioral therapy for insomnia
- Health education (Active Comparator): Health education group will attend online meeting, 1 hour weekly for 8 weeks.
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: cognitive behavioral therapy for insomnia — Online meeting, weekly for 8 weeks, to deliver CBTI by psychologist/ psychiatrist
  Arms: Cognitive behavioral therapy
Behavioral: Health education — Online meeting, weekly for 8 weeks, to deliver general health knowledge
  Arms: Health education

SUMMARY:
This study will explore the effects of cognitive behavioral therapy for insomnia (CBTI) compare to health educations in patients with type 2 diabetes (T2DM) with insomnia symptoms.

DETAILED DESCRIPTION:
This study will recruit participants with T2DM with insomnia symptoms and randomize them to weekly CBTI or health education for 8 weeks. Outcomes will be measured at baseline and 8 week, and 16 weeks (8 weeks post intervention).

Primary outcome will be subjective sleep quality as assessed by Pittsburgh Sleep Quality Index Secondary outcomes will be fasting glucose, hemoglobin A1C, insulin levels, high sensitivity c-reactive protein, objective sleep parameters from accelerometer, depressive symptoms, daytime sleepiness, quality of life, anxiety symptoms and stress symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus age 30 to 65 years old
* Hemoglobin A1C ≥ 6.5 but ≤ 10 %
* Have poor sleep quality as assessed by Insomnia Severity Index ≥ 15
* Receive the same hypoglycemic treatments 3 months before the intervention
* If using sleep aid, the dose needs to be stable for 3 months prior to the enrollment
* Ability to use the electronic devices (computer, tablet) and assess the internet
* Willing to attend all of the 8 sessions activities

Exclusion Criteria:

* Type 1 diabetes mellitus
* Night shift work
* Insulin therapy
* Severe hypoglycemia who required hospitalization or emergency department visit in the past 6 months
* History of diabetic ketoacidosis in the past 6 months
* Medically unstable conditions eg. renal replacement therapy, liver failure, heart failure, active cancer, epilepsy, unstable cerebrovascular disease
* Psychosis, uncontrolled depression
* Untreated obstructive sleep apnea or STOP-BANG ≥ 5
* Language/communication/hearing/sight disability
* Pregnancy or lactation
* Care giver of infant
* Harmful alcohol/smoking (≥15 standard-drink in men and ≥8 standard-drink in women)

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Subjective Sleep Quality | 16 weeks
  Subjective Sleep Quality as assessed by Pittsburgh Sleep Quality Index

SECONDARY OUTCOMES:
Metabolic parameters | 8 weeks
  Fasting glucose and insulin, hemoglobin A1C
High sensitivity c-reactive protein | 8 weeks
  serum sample for Hs-CRP
Patient reported outcomes | 16 weeks
  Questionnaires to assess depressive symptoms, stress, anxiety, daytime sleepiness, and quality of life
Objective sleep parameters | 8 weeks
  Sleep will be obtained using 1-week accelerometer recording

CONTACTS AND LOCATIONS:
Overall Officials: Similan Kirisri, Principal Investigator — Ramathibodi Hospital
Locations (1):
- Faculty of Medicine Ramathibodi Hospital Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No